CLINICAL TRIAL: NCT02065830
Title: ROBOticsSpinalCordInjuryEKSO: Outdoor and Indoor Mobility in People With SCI.
Brief Title: Safety Study of Outdoor and Indoor Mobility in People With Spinal Cord Injury (ROBOtics Spinal Cord Injury EKSO).
Acronym: ROBOSCIEKSO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROBOSCIEKSO
Record Dates: First submitted 2014-02-12; First posted 2014-02-19 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Spinal Cord Injury
Keywords: Robot; Spinal Cord Injury; Gait; Quality of life; Rehabilitation; Lower Limb
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robot Safety and Efficacy (Experimental): The subjects will undergo inpatient rehabilitation consisting of a treatment cycle of 30/40 training section using the robot EKSO system device, according to individually tailored exercise scheduling.
  The practice will include robot-assisted walking at variable speeds for 45/60 min and balance training.
  Interventions: Device: EKSO

INTERVENTIONS:
Device: EKSO — The subjects will undergo inpatient rehabilitation consisting of a treatment cycle of 30/40 training section using the robot EKSO system device, according to individually tailored exercise scheduling.
  The practice will include robot-assisted walking at variable speeds for 45/60 min and balance training.

SUMMARY:
The aim of this study will be to evaluate the safety and the efficacy of a new robotic exoskeleton device in subjects with Spinal Cord Injury (SCI) and in subjects with other neurological disease with an impairment of lower limbs.

DETAILED DESCRIPTION:
In this study, 30 participants with chronic spinal cord injury will undergo a 8-week training schedule for ambulation with the EKSO™ device.

Ekso™ is a wearable bionic suit which enables individuals with any amount of lower extremity weakness to stand up and walk over ground with a natural, full weight bearing, reciprocal gait. Walking is achieved by the user's weight shifts to activate sensors in the device which initiate steps. Battery-powered motors drive the legs, replacing deficient neuromuscular function.

Ekso provides functional based rehabilitation, over ground gait training, and upright, weight bearing exercise unlike any other. It has been designed for the needs of busy therapists treating a wide range of patients in a single day. The suit is strapped over the users´ clothing with easy adjustments to transition between patients in as little as five minutes.

Before, during and after training sessions the subjects will perform standardised assessments and complete questionnaires to assess the functional and psychological effects of the exoskeleton.

ELIGIBILITY:
Inclusion Criteria:

* Chronic motor complete or incomplete cervical and thoracic (C7-T12) spinal cord injury.
* Skin integrity.
* Adequate hip, knee and ankle range of motion.
* Spasticity level of 3 or less (Ashworth scale).

Exclusion Criteria:

* Cardiological or respiratory comorbidity.
* Hemodynamic instability.
* Presence of unhealed fractures.
* Presence of heterotopic ossification that may impede walking.
* Presence of osteoporosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Gait Spatiotemporal and Kinematic parameters at 6 months. | Ekso training at 0 and 8 weeks, and 24-week follow-up.
  Change in score between 0 and 24 weeks. 3D Gait Analysis will be collected at baseline (inclusion) (T0) after 30/40 robot session an expected average of 8 weeks (T1) and at the follow-up examination after 6 months from the training conclusion (T2).

SECONDARY OUTCOMES:
Participant Satisfaction Questionnaire. | Ekso training at 0 and 8 weeks, and 24-week follow-up
  Change in score between 0 and 24 weeks. The 10 questions will be asked for each subject during and upon the completion of the active participation phase of the treatment.
Change in blood pressure and heart rate during the training. | Ekso training at 0 and 8 weeks, and 24-week follow-up.
  Blood pressure and heart rate will be monitorized every day during the training and the data will be collected at baseline (inclusion) (T0) after 30/40 robot session an expected average of 8 weeks (T1) and at the follow-up examination after 6 months from the training conclusion (T2).
6 minutes walking test. | Ekso training at 0 and 8 weeks, and 24-week follow-up.
  Change in score between 0 and 24 weeks. The 6 minutes walking test will be collected in indoor and outdoor condition at baseline (inclusion) (T0) after 30/40 robot session an expected average of 8 weeks (T1) and at the follow-up examination after 6 months from the training conclusion (T2).
Timed Up and Go test. | Ekso training at 0 and 8 weeks, and 24-week follow-up.
  Change in score between 0 and 24 weeks. Timed Up and Go test will be collected in indoor and outdoor condition at baseline (inclusion) (T0) after 30/40 robot session an expected average of 8 weeks (T1) and at the follow-up examination after 6 months from the training conclusion (T2).

CONTACTS AND LOCATIONS:
Overall Officials: Patrizio Sale, MD, Principal Investigator — IRCCS San Raffaele Pisana Roma
Locations (2):
- Italy (2):
  - Fondazione Centri di Riabilitazione Padre Pio Onlus, San Giovanni Rotondo, Foggia
  - IRCCS San Raffaele Pisana Roma, Roma

REFERENCES:
- [Derived] Sale P, Russo EF, Russo M, Masiero S, Piccione F, Calabro RS, Filoni S. Effects on mobility training and de-adaptations in subjects with Spinal Cord Injury due to a Wearable Robot: a preliminary report. BMC Neurol. 2016 Jan 28;16:12. doi: 10.1186/s12883-016-0536-0. PMID 26818847